CLINICAL TRIAL: NCT01486979
Title: A Pharmacokinetic Randomized Study With a Parallel Group Design to Assess the Extent of Systemic Absorption of Estradiol During Treatment With a 10 µg or 25 µg Estradiol Vaginal Tablet Administered Once Daily for 2 Weeks Followed by 10 Weeks of Twice-Weekly Maintenance Therapy in Postmenopausal Women With Atrophic Vaginitis
Brief Title: Pharmacokinetic Assessment of the Absorption of Estradiol in Postmenopausal Women With Atrophic Vaginitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAG-1850; 2006-005957-31 (EudraCT Number)
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Menopause; Postmenopausal Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose (Experimental)
  Interventions: Drug: estradiol, 10 mcg
- High dose (Active Comparator)
  Interventions: Drug: estradiol, 25 mcg

INTERVENTIONS:
Drug: estradiol, 10 mcg — One vaginal tablet once daily in the morning during the first two weeks of treatment followed by one vaginal tablet twice weekly in the morning for 10 weeks
  Arms: Low dose
Drug: estradiol, 25 mcg — One vaginal tablet once daily in the morning during the first two weeks of treatment followed by one vaginal tablet twice weekly in the morning for 10 weeks
  Arms: High dose

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to to evaluate the extent of systemic absorption of estradiol during treatment with two different doses of estradiol in postmenopausal women with atrophic vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to use German language in speaking and writing
* Postmenopausal women with at least 5 years after last menstruation, or bilateral oophorectomy performed two years or more prior to the time of screening
* Serum FSH (Follicle Stimulating Hormone) levels above 40 mIU/ml and estradiol below 20 pg/ml
* Maximum 5% superficial cells as assessed by evaluation of vaginal cytology
* Endometrial thickness below 4.0 mm (double layer), as measured by transvaginal ultrasound (if applicable)
* Availability of a normal mammogram within one year prior to trial start
* Good general health as assessed by the Investigator and based on medical history, and physical and laboratory examinations

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Known, suspected or past history of breast cancer
* Known, suspected or past estrogen dependent neoplasia e.g. endometrial cancer
* Endometrial hyperplasia or endometrial polyps diagnosed during the screening period
* Abnormal genital bleeding of unknown etiology
* Previous estrogen and/ or progestin hormone replacement therapy

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC)

SECONDARY OUTCOMES:
Average plasma concentration (C average)
Maximal concentration (Cmax)
Minimal concentration (Cmin)
Time of maximal concentration (tmax)
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neu-Ulm, Germany

REFERENCES:
- [Result] Eugster-Hausmann M, Waitzinger J, Lehnick D. Minimized estradiol absorption with ultra-low-dose 10 microg 17beta-estradiol vaginal tablets. Climacteric. 2010 Jun;13(3):219-27. doi: 10.3109/13697137.2010.483297. PMID 20423242
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com